CLINICAL TRIAL: NCT01140100
Title: A Comparative Study of Depth of Anesthesia Monitored by BIS Values in Two Anesthesia Techniques
Brief Title: A Comparative Study of Depth of Anesthesia Monitored by Bispectral Index (BIS) Values
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 85-3211
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2007-01

CONDITIONS: Anesthetics
MeSH Terms: interventions — Propofol; Thiopental

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol-propofol (Active Comparator)
  Interventions: Drug: propofol
- thiopental-propofol (Experimental)
  Interventions: Drug: thiopental,propofol

INTERVENTIONS:
Drug: propofol
  Arms: propofol-propofol
Drug: thiopental,propofol
  Arms: thiopental-propofol

SUMMARY:
The aim of this study is to determine whether induction of anesthesia with thiopental followed by propofol infusion is able to maintain sufficient depth of anesthesia .

ELIGIBILITY:
Inclusion Criteria:

* being adult
* having ASA I or II
* scheduled for elective cataract surgery under general anesthesia

Exclusion Criteria:

* massive obesity
* intake of any central nervous system (CNS) stimulants
* intake of CNS depressants
* intake of Tricyclic antidepressants
* known adverse reaction to the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sina Ghaffaripour, M.D, Principal Investigator — Shiraz University of Medical Sciences; Hilda Mahmoudi, M.D, Study Director — Shiraz University of Medical Sciences
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran